CLINICAL TRIAL: NCT04229264
Title: Efficacy and Safety of Apixaban in Reducing Restenosis and Limb Loss in Subjects With Symptomatic Peripheral Artery Disease (PAD) Undergoing Infrapopliteal Endovascular Peripheral Revascularization Procedures in Patients With Critical Limb
Brief Title: Efficacy and Safety of Apixaban in Reducing Restenosis and Limb Loss in PAD Patients.
Acronym: AGRIPPA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Science Valley Research Institute (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGRIPPA/EMRISTA 2018
Record Dates: First submitted 2019-12-10; First posted 2020-01-18 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Critical Limb Ischemia
Keywords: Post-infrapopliteal angioplasty
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — apixaban; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Aspirin 100 mg (oral, once-daily) for 1 year plus Clopidogrel 75 mg (oral, once-daily) for 3 months.
  Interventions: Drug: ASA; Drug: Clopidogrel 75mg
- Apixaban group (Experimental): Apixaban 2.5 mg (oral, twice daily) for 1 year plus Aspirin 100 mg (oral, once-daily) for 1 year.
  Interventions: Drug: Apixaban; Drug: ASA

INTERVENTIONS:
Drug: Apixaban — Oral Apixaban 2.5 mg twice daily for one year
  Other Names: Doppler Ultrasound Follow-up 1, 3, 6 and 12 months
  Arms: Apixaban group
Drug: ASA — Acetil Salicilic Acid 100mg once daily for one year
Drug: Clopidogrel 75mg — Clopidogrel 75mg once daily for 3 months
  Other Names: Doppler Ultrasound Follow-up 1, 3, 6 and 12 months
  Arms: Control group

SUMMARY:
This study will evaluate the efficacy and safety of apixaban 2.5 mg twice daily plus aspirin compared to the standard treatment (clopidogrel plus aspirin) in patients with critical limb ischemia undergoing infrapopliteal arterial endovascular intervention.

DETAILED DESCRIPTION:
This study is a multicentre, parallel-group, prospective, randomized open-label, blinded-endpoint adjudication, proof-of-concept, and exploratory trial. Two hundred patients will be randomized in a 1:1 ratio, 72 hours after successful infrapopliteal angioplasty for critical limb ischemia. In the study group, patients will receive oral apixaban 2.5mg twice daily plus aspirin 100 mg once-daily for 12 months. In the control group, aspirin 100 mg once-daily will be taken for 1 year on a background of clopidogrel (75mg daily) for the first three months. The primary endpoint is the composite of target lesion revascularization (TLR), major amputation or restenosis/occlusion (RAS) plus MACE (myocardial infarction, stroke, and cardiovascular death) at 12 months. The primary safety endpoint is the composite of major bleeding and clinically relevant non-major bleeding at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Age>18 years old.
* Negative serum pregnancy test (in women of childbearing only).
* Patients submitted to endovascular procedures below-the-knee by not exclusively.
* Patient understands and is willing and able to comply with the study instructions and follow-up visit.
* More than 70% stenosis or occlusion of the three distal arteries including or not the tibiofibular trunk (TFT).
* Tissue loss (Rutherford 5).
* One or more patent vessel of pedal arch.

Exclusion Criteria:

* TASC II D femoral and/or popliteal occlusion.
* Life expectancy less than 1 year.
* Allergy or contraindication to apixaban treatment.
* Allergy or contraindication to dual antiplatelet treatment.
* Creatinine clearance less than 30mL/min.
* Planned major amputation before procedure.
* Hybrid procedure (open and endovascular).
* Use of fibrinolytic in the past 10 days.
* Known HIV infection.
* Liver disease (acute or chronic hepatitis and cirrhosis).
* Drug addiction or alcohol abuse 12 months before the randomization.
* Concomitant medications thatinhibit the CYP 3A4 cytochrome and P glycoprotein (ketoconazole, Iitraconazole, ritonavir).
* Platelets count inferior to 100x109/L.
* INR more than 1.5.
* History or condition with high risk of bleeding: Eg. Trauma within 30 days before randomization, gastrointestinal bleeding 6 month before the randomization, intra-ocular, spinal, intra-articular bleeding (any time before), AV malformation, cerebral aneurysm and hypertension without control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2022-02-02 (Estimated); Study Completion 2022-05-02 (Estimated)

PRIMARY OUTCOMES:
Restenosis of the treated infrapopliteal artery | 12 months
  Number of patients with absence of flow or >2.4 sistolic index obtained by Duplex Scan
Major amputation | 12 months
  Number of patients who underwent amputation of the leg above the ankle
Clinical driven-target lesion revascularization | 12 months
  Number of patients who was submitted by reintervention of the treated infrapopliteal artery based on the clinical status
Major cardiovascular events | 12 months
  Number of patients who present one of those: myocardial infarction, stroke and cardiovascular death

SECONDARY OUTCOMES:
Bleeding | 12 months
  Number of patients who present major bleeding (MB) or clinically relevant non-major bleeding, using the ISTH criteria
Healing | 12 months
  Time to total healing measured by the Imitomeasure program.

CONTACTS AND LOCATIONS:
Locations (1):
- IAMSPE - Sao Paulo Public Servants Hospital, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferraresi R, Centola M, Ferlini M, Da Ros R, Caravaggi C, Assaloni R, Sganzaroli A, Pomidossi G, Bonanomi C, Danzi GB. Long-term outcomes after angioplasty of isolated, below-the-knee arteries in diabetic patients with critical limb ischaemia. Eur J Vasc Endovasc Surg. 2009 Mar;37(3):336-42. doi: 10.1016/j.ejvs.2008.12.001. Epub 2008 Dec 27. PMID 19112033
- [Background] Tsetis D, Belli AM. The role of infrapopliteal angioplasty. Br J Radiol. 2004 Dec;77(924):1007-15. doi: 10.1259/bjr/97382129. PMID 15569642
- [Background] Shishehbor MH, Hammad TA, Zeller T, Baumgartner I, Scheinert D, Rocha-Singh KJ. An analysis of IN.PACT DEEP randomized trial on the limitations of the societal guidelines-recommended hemodynamic parameters to diagnose critical limb ischemia. J Vasc Surg. 2016 May;63(5):1311-7. doi: 10.1016/j.jvs.2015.11.042. Epub 2016 Feb 6. PMID 26860642
- [Background] El-Sayed H, Bennett ME, Loh TM, Davies MG. Retrograde Pedal Access and Endovascular Revascularization: A Safe and Effective Technique for High-Risk Patients with Complex Tibial Vessel Disease. Ann Vasc Surg. 2016 Feb;31:91-8. doi: 10.1016/j.avsg.2015.09.015. Epub 2015 Nov 26. PMID 26627317
- [Background] Wu R, Yao C, Wang S, Xu X, Wang M, Li Z, Wang S. Percutaneous transluminal angioplasty versus primary stenting in infrapopliteal arterial disease: a meta-analysis of randomized trials. J Vasc Surg. 2014 Jun;59(6):1711-20. doi: 10.1016/j.jvs.2014.03.012. PMID 24836770
- [Background] Silingardi R, Tasselli S, Cataldi V, Moratto R, Gennai S, Coppi G, Marcheselli L, Coppi G. Bifurcated coronary stents for infrapopliteal angioplasty in critical limb ischemia. J Vasc Surg. 2013 Apr;57(4):1006-13. doi: 10.1016/j.jvs.2012.09.080. Epub 2013 Jan 21. PMID 23343667
- [Background] Gutzeit A, Schoch E, Sautter T, Jenelten R, Graf N, Binkert CA. Antegrade access to the superficial femoral artery with ultrasound guidance: feasibility and safety. J Vasc Interv Radiol. 2010 Oct;21(10):1495-500. doi: 10.1016/j.jvir.2010.03.021. PMID 20801678
- [Background] Marcus AJ, Lotzof K, Howard A. Access to the superficial femoral artery in the presence of a "hostile groin": a prospective study. Cardiovasc Intervent Radiol. 2007 May-Jun;30(3):351-4. doi: 10.1007/s00270-005-0347-y. PMID 17295080
- [Background] Liistro F, Porto I, Angioli P, Grotti S, Ricci L, Ducci K, Falsini G, Ventoruzzo G, Turini F, Bellandi G, Bolognese L. Drug-eluting balloon in peripheral intervention for below the knee angioplasty evaluation (DEBATE-BTK): a randomized trial in diabetic patients with critical limb ischemia. Circulation. 2013 Aug 6;128(6):615-21. doi: 10.1161/CIRCULATIONAHA.113.001811. PMID 23797811
- [Background] Adam DJ, Beard JD, Cleveland T, Bell J, Bradbury AW, Forbes JF, Fowkes FG, Gillepsie I, Ruckley CV, Raab G, Storkey H; BASIL trial participants. Bypass versus angioplasty in severe ischaemia of the leg (BASIL): multicentre, randomised controlled trial. Lancet. 2005 Dec 3;366(9501):1925-34. doi: 10.1016/S0140-6736(05)67704-5. PMID 16325694
- [Background] Romiti M, Albers M, Brochado-Neto FC, Durazzo AE, Pereira CA, De Luccia N. Meta-analysis of infrapopliteal angioplasty for chronic critical limb ischemia. J Vasc Surg. 2008 May;47(5):975-981. doi: 10.1016/j.jvs.2008.01.005. Epub 2008 Apr 18. PMID 18372148
- [Background] Faglia E, Dalla Paola L, Clerici G, Clerissi J, Graziani L, Fusaro M, Gabrielli L, Losa S, Stella A, Gargiulo M, Mantero M, Caminiti M, Ninkovic S, Curci V, Morabito A. Peripheral angioplasty as the first-choice revascularization procedure in diabetic patients with critical limb ischemia: prospective study of 993 consecutive patients hospitalized and followed between 1999 and 2003. Eur J Vasc Endovasc Surg. 2005 Jun;29(6):620-7. doi: 10.1016/j.ejvs.2005.02.035. Epub 2005 Mar 28. PMID 15878541
- [Background] Nair V, Chaisson G, Abben R. Strategies in infrapopliteal intervention: improving outcomes in challenging patients. J Interv Cardiol. 2009 Feb;22(1):27-36. doi: 10.1111/j.1540-8183.2008.00412.x. No abstract available. PMID 19281520
- [Background] Sumpio BE, Forsythe RO, Ziegler KR, van Baal JG, Lepantalo MJ, Hinchliffe RJ. Clinical implications of the angiosome model in peripheral vascular disease. J Vasc Surg. 2013 Sep;58(3):814-26. doi: 10.1016/j.jvs.2013.06.056. PMID 23972249
- [Background] Sadaghianloo N, Jean-Baptiste E, Declemy S, Mousnier A, Brizzi S, Hassen-Khodja R. Percutaneous angioplasty of long tibial occlusions in critical limb ischemia. Ann Vasc Surg. 2013 Oct;27(7):894-903. doi: 10.1016/j.avsg.2013.02.008. PMID 23993107
- [Background] Singh GD, Armstrong EJ, Yeo KK, Singh S, Westin GG, Pevec WC, Dawson DL, Laird JR. Endovascular recanalization of infrapopliteal occlusions in patients with critical limb ischemia. J Vasc Surg. 2014 May;59(5):1300-7. doi: 10.1016/j.jvs.2013.11.061. Epub 2014 Jan 3. PMID 24393279
- [Background] Saqib NU, Domenick N, Cho JS, Marone L, Leers S, Makaroun MS, Chaer RA. Predictors and outcomes of restenosis following tibial artery endovascular interventions for critical limb ischemia. J Vasc Surg. 2013 Mar;57(3):692-9. doi: 10.1016/j.jvs.2012.08.115. Epub 2013 Jan 23. PMID 23351646
- [Background] Scheinert D, Ulrich M, Scheinert S, Sax J, Braunlich S, Biamino G. Comparison of sirolimus-eluting vs. bare-metal stents for the treatment of infrapopliteal obstructions. EuroIntervention. 2006 Aug;2(2):169-74. PMID 19755256
- [Background] Silingardi R, Lauricella A, Coppi G, Chester J, Trevisi-Borsari G, Corvi V, Marcheselli L, Coppi G. Durability and efficacy of tibial arterial stent placement for critical limb ischemia. J Vasc Interv Radiol. 2015 Apr;26(4):475-83.e2. doi: 10.1016/j.jvir.2014.11.044. Epub 2015 Feb 7. PMID 25666627
- [Background] Ozkan U, Oguzkurt L, Tercan F. Atherosclerotic risk factors and segmental distribution in symptomatic peripheral artery disease. J Vasc Interv Radiol. 2009 Apr;20(4):437-41. doi: 10.1016/j.jvir.2009.01.010. PMID 19328423
- [Background] Bolia A, Brennan J, Bell PR. Recanalisation of femoro-popliteal occlusions: improving success rate by subintimal recanalisation. Clin Radiol. 1989 May;40(3):325. doi: 10.1016/s0009-9260(89)80231-4. No abstract available. PMID 2526702
- [Background] Dormandy JA, Rutherford RB. Management of peripheral arterial disease (PAD). TASC Working Group. TransAtlantic Inter-Society Consensus (TASC). J Vasc Surg. 2000 Jan;31(1 Pt 2):S1-S296. No abstract available. PMID 10666287
- [Background] Kawarada O, Yokoi Y, Higashimori A, Waratani N, Waseda K, Honda Y, Fitzgerald PJ. Stent-assisted below-the-ankle angioplasty for limb salvage. J Endovasc Ther. 2011 Feb;18(1):32-42. doi: 10.1583/10-3214.1. PMID 21314346
- [Background] Kawarada O, Yasuda S, Nishimura K, Sakamoto S, Noguchi M, Takahi Y, Harada K, Ishihara M, Ogawa H. Effect of single tibial artery revascularization on microcirculation in the setting of critical limb ischemia. Circ Cardiovasc Interv. 2014 Oct;7(5):684-91. doi: 10.1161/CIRCINTERVENTIONS.113.001311. Epub 2014 Aug 19. PMID 25138035
- [Background] Peeters Weem SM, van Haelst ST, den Ruijter HM, Moll FL, de Borst GJ. Lack of Evidence for Dual Antiplatelet Therapy after Endovascular Arterial Procedures: A Meta-analysis. Eur J Vasc Endovasc Surg. 2016 Aug;52(2):253-62. doi: 10.1016/j.ejvs.2016.04.023. Epub 2016 May 27. PMID 27241270
- [Background] Hirsch AT, Haskal ZJ, Hertzer NR, Bakal CW, Creager MA, Halperin JL, Hiratzka LF, Murphy WR, Olin JW, Puschett JB, Rosenfield KA, Sacks D, Stanley JC, Taylor LM Jr, White CJ, White J, White RA, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Hunt SA, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American Association for Vascular Surgery; Society for Vascular Surgery; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine and Biology; Society of Interventional Radiology; ACC/AHA Task Force on Practice Guidelines Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease; American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; Vascular Disease Foundation. ACC/AHA 2005 Practice Guidelines for the management of patients with peripheral arterial disease (lower extremity, renal, mesenteric, and abdominal aortic): a collaborative report from the American Association for Vascular Surgery/Society for Vascular Surgery, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, Society of Interventional Radiology, and the ACC/AHA Task Force on Practice Guidelines (Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease): endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; and Vascular Disease Foundation. Circulation. 2006 Mar 21;113(11):e463-654. doi: 10.1161/CIRCULATIONAHA.106.174526. No abstract available. PMID 16549646
- [Background] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). J Vasc Surg. 2007 Jan;45 Suppl S:S5-67. doi: 10.1016/j.jvs.2006.12.037. No abstract available. PMID 17223489
- [Background] Alonso-Coello P, Bellmunt S, McGorrian C, Anand SS, Guzman R, Criqui MH, Akl EA, Vandvik PO, Lansberg MG, Guyatt GH, Spencer FA. Antithrombotic therapy in peripheral artery disease: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e669S-e690S. doi: 10.1378/chest.11-2307. PMID 22315275
- [Background] European Stroke Organisation; Tendera M, Aboyans V, Bartelink ML, Baumgartner I, Clement D, Collet JP, Cremonesi A, De Carlo M, Erbel R, Fowkes FG, Heras M, Kownator S, Minar E, Ostergren J, Poldermans D, Riambau V, Roffi M, Rother J, Sievert H, van Sambeek M, Zeller T; ESC Committee for Practice Guidelines. ESC Guidelines on the diagnosis and treatment of peripheral artery diseases: Document covering atherosclerotic disease of extracranial carotid and vertebral, mesenteric, renal, upper and lower extremity arteries: the Task Force on the Diagnosis and Treatment of Peripheral Artery Diseases of the European Society of Cardiology (ESC). Eur Heart J. 2011 Nov;32(22):2851-906. doi: 10.1093/eurheartj/ehr211. Epub 2011 Aug 26. No abstract available. PMID 21873417
- [Background] Yen HT, Hsieh MJ, Wu CC, Lee FY. Effect of systemic urokinase infusion after lower limb percutaneous transluminal angioplasty on limb salvage rate in patients with late-stage critical limb ischemia. Eur J Vasc Endovasc Surg. 2014 Oct;48(4):414-22. doi: 10.1016/j.ejvs.2014.04.006. Epub 2014 Jun 28. PMID 24984839
- [Background] Dosluoglu HH, Harris LM. Endovascular management of subacute lower extremity ischemia. Semin Vasc Surg. 2008 Dec;21(4):167-79. doi: 10.1053/j.semvascsurg.2008.11.002. PMID 19073306
- [Background] Lam RC, Shah S, Faries PL, McKinsey JF, Kent KC, Morrissey NJ. Incidence and clinical significance of distal embolization during percutaneous interventions involving the superficial femoral artery. J Vasc Surg. 2007 Dec;46(6):1155-9. doi: 10.1016/j.jvs.2007.07.058. PMID 18154991
- [Background] Motarjeme A, Gordon GI, Bodenhagen K. Thrombolysis and angioplasty of chronic iliac artery occlusions. J Vasc Interv Radiol. 1995 Nov-Dec;6(6 Pt 2 Suppl):66S-72S. doi: 10.1016/s1051-0443(95)71251-9. PMID 8770845
- [Background] Wholey MH, Maynar MA, Wholey MH, Pulido-Duque JM, Reyes R, Jarmolowski CR, Castaneda WR. Comparison of thrombolytic therapy of lower-extremity acute, subacute, and chronic arterial occlusions. Cathet Cardiovasc Diagn. 1998 Jun;44(2):159-69. doi: 10.1002/(sici)1097-0304(199806)44:23.0.co;2-5. PMID 9637438
- [Background] Lee HF, Chan YH, Wang CL. Using Rivaroxaban as Thrombolytic Treatment for a Patient of Pedal Arch Arterial Thrombosis with Suboptimal Result of Endovascular Therapy. Acta Cardiol Sin. 2016 Sep;32(5):623-626. doi: 10.6515/acs20151229a. PMID 27713614
- [Background] Undas A, Ariens RA. Fibrin clot structure and function: a role in the pathophysiology of arterial and venous thromboembolic diseases. Arterioscler Thromb Vasc Biol. 2011 Dec;31(12):e88-99. doi: 10.1161/ATVBAHA.111.230631. Epub 2011 Aug 11. PMID 21836064
- [Background] Warfarin Antiplatelet Vascular Evaluation Trial Investigators; Anand S, Yusuf S, Xie C, Pogue J, Eikelboom J, Budaj A, Sussex B, Liu L, Guzman R, Cina C, Crowell R, Keltai M, Gosselin G. Oral anticoagulant and antiplatelet therapy and peripheral arterial disease. N Engl J Med. 2007 Jul 19;357(3):217-27. doi: 10.1056/NEJMoa065959. PMID 17634457
- [Background] Greig SL, Garnock-Jones KP. Apixaban: A Review in Venous Thromboembolism. Drugs. 2016 Oct;76(15):1493-1504. doi: 10.1007/s40265-016-0644-6. PMID 27653758
- [Background] Beyer-Westendorf J, Lensing AW, Arya R, Bounameaux H, Cohen AT, Wells PS, Middeldorp S, Verhamme P, Hughes R, Kucher N, Pap AF, Trajanovic M, Prins MH, Prandoni P, Weitz JI. Choosing wisely: The impact of patient selection on efficacy and safety outcomes in the EINSTEIN-DVT/PE and AMPLIFY trials. Thromb Res. 2017 Jan;149:29-37. doi: 10.1016/j.thromres.2016.11.014. Epub 2016 Nov 21. PMID 27886530
- [Background] Bleker SM, Cohen AT, Buller HR, Agnelli G, Gallus AS, Raskob GE, Weitz JI, Curto M, Sisson M, Middeldorp S. Clinical presentation and course of bleeding events in patients with venous thromboembolism, treated with apixaban or enoxaparin and warfarin. Results from the AMPLIFY trial. Thromb Haemost. 2016 Nov 30;116(6):1159-1164. doi: 10.1160/TH16-02-0137. Epub 2016 Sep 1. PMID 27583312
- [Background] Blomback M, He S, Bark N, Wallen HN, Elg M. Effects on fibrin network porosity of anticoagulants with different modes of action and reversal by activated coagulation factor concentrate. Br J Haematol. 2011 Mar;152(6):758-65. doi: 10.1111/j.1365-2141.2010.08546.x. Epub 2011 Jan 20. PMID 21250974
- [Background] Stoner MC, Calligaro KD, Chaer RA, Dietzek AM, Farber A, Guzman RJ, Hamdan AD, Landry GJ, Yamaguchi DJ; Society for Vascular Surgery. Reporting standards of the Society for Vascular Surgery for endovascular treatment of chronic lower extremity peripheral artery disease. J Vasc Surg. 2016 Jul;64(1):e1-e21. doi: 10.1016/j.jvs.2016.03.420. PMID 27345516
- [Background] Siablis D, Karnabatidis D, Katsanos K, Kagadis GC, Kraniotis P, Diamantopoulos A, Tsolakis J. Sirolimus-eluting versus bare stents after suboptimal infrapopliteal angioplasty for critical limb ischemia: enduring 1-year angiographic and clinical benefit. J Endovasc Ther. 2007 Apr;14(2):241-50. doi: 10.1177/152660280701400217. PMID 17484536
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Mills JL Sr, Conte MS, Armstrong DG, Pomposelli FB, Schanzer A, Sidawy AN, Andros G; Society for Vascular Surgery Lower Extremity Guidelines Committee. The Society for Vascular Surgery Lower Extremity Threatened Limb Classification System: risk stratification based on wound, ischemia, and foot infection (WIfI). J Vasc Surg. 2014 Jan;59(1):220-34.e1-2. doi: 10.1016/j.jvs.2013.08.003. Epub 2013 Oct 12. PMID 24126108
- [Background] Bollinger A, Breddin K, Hess H, Heystraten FM, Kollath J, Konttila A, Pouliadis G, Marshall M, Mey T, Mietaschk A, Roth FJ, Schoop W. Semiquantitative assessment of lower limb atherosclerosis from routine angiographic images. Atherosclerosis. 1981 Feb-Mar;38(3-4):339-46. doi: 10.1016/0021-9150(81)90050-2. PMID 7225173
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2011;9(8):672-7. doi: 10.1016/j.ijsu.2011.09.004. Epub 2011 Oct 13. No abstract available. PMID 22019563
- [Background] Avezum A, Lopes RD, Schulte PJ, Lanas F, Gersh BJ, Hanna M, Pais P, Erol C, Diaz R, Bahit MC, Bartunek J, De Caterina R, Goto S, Ruzyllo W, Zhu J, Granger CB, Alexander JH. Apixaban in Comparison With Warfarin in Patients With Atrial Fibrillation and Valvular Heart Disease: Findings From the Apixaban for Reduction in Stroke and Other Thromboembolic Events in Atrial Fibrillation (ARISTOTLE) Trial. Circulation. 2015 Aug 25;132(8):624-32. doi: 10.1161/CIRCULATIONAHA.114.014807. Epub 2015 Jun 23. PMID 26106009
- [Background] Agnelli G, Buller HR, Cohen A, Curto M, Gallus AS, Johnson M, Masiukiewicz U, Pak R, Thompson J, Raskob GE, Weitz JI; AMPLIFY Investigators. Oral apixaban for the treatment of acute venous thromboembolism. N Engl J Med. 2013 Aug 29;369(9):799-808. doi: 10.1056/NEJMoa1302507. Epub 2013 Jul 1. PMID 23808982
- [Background] Biagioni RB, Biagioni LC, Nasser F, Burihan MC, Ingrund JC, Neser A, Miranda F Jr. Infrapopliteal Angioplasty of One or More than One Artery for Critical Limb Ischaemia: A Randomised Clinical Trial. Eur J Vasc Endovasc Surg. 2018 Apr;55(4):518-527. doi: 10.1016/j.ejvs.2017.12.022. PMID 29402670
- [Derived] Biagioni RB, Lopes RD, Agati LB, Sacilotto R, Wolosker N, Sobreira ML, de Freitas Soares BL, Joviliano EE, Bernardi WH, Junior VC, Caffaro RA, Fioranelli A, Van Bellen B, Casella IB, Fidelis RJR, Flumignan RLG, Comerota AJ, Ramacciotti E. Rationale and design for the study Apixaban versus ClopidoGRel on a background of aspirin in patient undergoing InfraPoPliteal angioplasty for critical limb ischemia: AGRIPPA trial. Am Heart J. 2020 Sep;227:100-106. doi: 10.1016/j.ahj.2020.06.010. Epub 2020 Jun 23. PMID 32730905